CLINICAL TRIAL: NCT04006496
Title: Expressive Writing to Address Distress in Hospitalized Adults With Acute Myeloid Leukemia (AML): a Pilot Randomized Clinical Trial
Brief Title: AML Expressive Writing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment issues due to COVID-19 pandemic.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00100520
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention (Experimental): In-patient, Chemotherapy patients in this arm will receive the expressive writing intervention twice each week for two weeks. These writing samples will be reviewed and analyzed. These patients will receive coaching from an expert expressive writing coach and will be allowed to ask questions and receive guidance. All patients will receive standard of care treatment in addition to the intervention.
  Interventions: Behavioral: Expressive Writing Coaching
- Control (No Intervention): Patients in the control group will not interface with the expressive writing coach for guidance nor have their writing samples reviewed and analyzed. All patients in the control arm will still receive standard care

INTERVENTIONS:
Behavioral: Expressive Writing Coaching — For the intervention group, a trained expressive writing expert/coach will introduce the expressive writing concept to consented patients during the first visit, followed by an introduction of the first expressive writing exercise and prompt. The expert/coach will introduce new writing prompts at each subsequent visit. A script containing each visit's writing prompt and instructions will also be left with the patients for future use and/or reference. The trained clinician will collect, read, and analyze the writing sample using a health coaching technique by: 1) summarizing what the patient wrote, 2) evoking double-sided reflection by reading back the writing sample to the patient, and 3) developing a metaphor and review with the patient. Patients will also have the opportunity to ask the trained clinician questions and receive guidance.
  Arms: Experimental: Intervention

SUMMARY:
A randomized, pilot feasibility and preliminary efficacy study to test such an intervention among hospitalized patients with AML who are receiving high-dose chemotherapy. Subjects randomized to the intervention arm will participate in a total of four, separate 1-hour expressive writing sessions that include the delivery of writing prompts, instructions, writing analyses, and coaching from a trained facilitator, delivered over the course of 2 weeks. Subjects randomized to the control arm of the study will receive standard care plus neutral writing prompts and instructions, but writing analyses and coaching from a trained facilitator will not be provided.

DETAILED DESCRIPTION:
To determine the feasibility, acceptability, and preliminary efficacy of an expressive writing intervention in this population, the investigators will recruit a total of 30 AML patients (15 patients in each study arm) at time of admission to Duke University Hospital for initiation of inpatient chemotherapy. To ensure homogeneity among enrolled patients, the investigators will restrict enrollment to within a 4-day window after starting chemotherapy. Although the investigators anticipate little attrition since patients are hospitalized for the entirety of the intervention, some may discontinue the study due to becoming critically ill. The investigators will thus recruit 30 patients in the event of 25% attrition to still meet the goal of at least 10 evaluable patients completing the study in each study arm.

To begin the study, patients will complete baseline surveys including demographics, consisting of the following:

* Conner-Davidson Resilience Scale (CD-RISC)21 • Patient Health Questionnaire-8 (PHQ-8)22
* Generalized Anxiety Disorder 7-item (GAD-7)23 • FACT-Leu quality of life scale for leukemia24
* Rumination Response Scale (RRS)25 • Demographics

Patients will receive the expressive writing intervention twice each week for two weeks for a total of four sessions. For the intervention group (n=15), Dr. Evans (co-investigator and trained expressive writing expert/coach) will introduce the expressive writing concept to consented patients during the first visit, followed by an introduction of the first expressive writing exercise and prompt. Dr. Evans will introduce new writing prompts at each subsequent visit. A script containing each visit's writing prompt and instructions will also be left with the patients for future use and/or reference. The trained clinician will collect, read, and analyze the writing sample using a health coaching technique by: 1) summarizing what the patient wrote, 2) evoking double-sided reflection by reading back the writing sample to the patient, and 3) developing a metaphor and review with the patient. Patients will also have the opportunity to ask the trained clinician questions and receive guidance. Patients consented and randomized into the control group (n=15) will receive the writing prompts with instructions for use from the research study coordinator. Patients in the control group will not interface with the interventionist, nor have their writing samples reviewed and analyzed. The control group will also not receive coaching regarding their writing samples from the interventionist, but the research study coordinator will collect the patients' writing samples at each of the four visits. Of note is that all patients will still receive standard care that includes attention to psychological distress by nursing staff and by physicians and advanced practice clinicians, as well as recreational therapy services, social work services, and available stress management services at the request of the primary cancer care team on the 9100 inpatient ward. After two weeks, participants will complete the same surveys as listed above (except demographics), as well as follow-up assessments at 4-weeks and 3-months.

The expressive writing prompts will consist of six modules containing the following expressive writing prompts:

1. Introduction to Expressive Writing and Transactional Writing Prompt
2. Personal Story about Your Experience with Cancer
3. Your Cancer form the Perspective of a Different Person
4. Legacy Writing Prompt
5. Mindful Writing Prompt
6. Closure Instructions to Encourage Continuing Expressive Writing

ELIGIBILITY:
Inclusion Criteria:

* At least age 18
* Capacity to give consent
* Diagnosis of acute myeloid leukemia (AML)
* Fluent in English
* Starting a new line of in-patient chemotherapy at Duke (in the last 4 days)

Exclusion Criteria:

* Patients too sick to participate per clinician discretion
* Patients that are not able to read or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Priori | 4 weeks
  The proportion of enrolled subjects who complete the study (including completing all writing tasks/coaching visits, and completing the surveys). The primary endpoint will be met if at least 80% of enrolled subjects do so.

SECONDARY OUTCOMES:
Change in resilience | Baseline, 4 weeks
  Change in Resilience based on Connor-Davidson Resilience 10-Item, 5-point scale (0-4), with higher scores reflecting greater resilience.
Change in depressive symptoms | Baseline, 4 weeks
  Measurements in depression and depressive symptoms based on Patient Health Questionnaire-8 (8-Item diagnostic instrument).
Change in patient's mental health status | Baseline, 4 weeks
  Change in patient's mental health status based on Generalized Anxiety Disorder (GAD-) (7-Item, self-report anxiety questionnaire).
Changes in cancer-related quality of life: Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu) (44-Item, 5-level Likert scale | Baseline, 4 weeks
  Assessment of cancer-related quality of life, with a specific subscale emphasizing concerns common among patients with leukemias using the Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu) (44-Item, 5-level Likert scale.
Measurement of brooding and reflective pondering | 4 weeks
  Measurement of two aspects of rumination using Rumination Response Scale (RRS) (22-Item, 4-Point scale: 1-Almost Never, 2-Sometimes, 3-Often, 4- Almost always, Level Likert Scale instrument)
Measurement of aspects of mood, intensity of expressions, and value and meaning. | 4 weeks
  Aspects of mood, intensity of expressions, and value and meaning will be measured using the Post Writing Reflection Survey (PWR) (5-Item, 10-Point scale (0-10), where 0= Not at All and 10= A Great Deal)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas LeBlanc, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No